CLINICAL TRIAL: NCT04089774
Title: Comparison of the Benefit Experienced by Patients With Ankylosing Spondylitis, Under Biotherapy, During Management by an Adapted Physical Activity Compared to a Standard Treatment by Kinesitherapy.
Brief Title: Benefit of Adapted Physical Activity for Patients Suffering From Ankylosing Spondylitis
Acronym: SPIKE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Denis Arniaud, principal investigator, Rheumatology department head, Hospital St. Joseph, Marseille, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ID RCB 2019-A00138-49
Record Dates: First submitted 2019-06-26; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity (APA) (Experimental): Supported by an Adapted Physical Activity (APA), at the rate of 3 sessions per week supervised by the association SCO STE MARGUERITE, spread over 12 months
  Interventions: Behavioral: Adapted Physical Activity (APA)
- Kiné (No Intervention): Standard physiotherapy treatment, at least 20 sessions, renewed at least once, spread over 12 months

INTERVENTIONS:
Behavioral: Adapted Physical Activity (APA) — Supported by an Adapted Physical Activity (APA), at the rate of 3 sessions per week supervised by the association SCO STE MARGUERITE, spread over 12 months
  Arms: Adapted Physical Activity (APA)

SUMMARY:
The current management of Spondylarthritis Ankylosant (SA), according to the recommendations of the HAS (High Authority of Health), must be a multidisciplinary global approach coordinated by the rheumatologist combining a pharmacological aspect (NSAID, analgesics, biotherapy ...) and not pharmacological (physical treatments, educational approaches, social measures ...). The therapeutic aim of this management is to achieve a low level of activity of the disease and a decrease of the repercussion of this one in the daily life of the patient.

The standard physical treatment currently provided is physiotherapy. This can be prescribed throughout the disease by the rheumatologist, adapted to the stage of AS and the clinical condition of the patient. The medical teams note in their daily practice that there may be a lack of attendance of patients at prescribed physiotherapy sessions. This has been confirmed in research on certain chronic rheumatic diseases, including AS, for which patients became less adherent to physical treatments and thus lost the expected benefits, particularly in terms of the functional impact of AS in the patient's daily life. (BASFI). Various studies have also shown that combining several physical activities (including aerobic and muscle building) or / and performing them in groups at a regular frequency (three times a week) could significantly improve several AS parameters, including BASFI.

From these different findings, we hypothesized that a multidisciplinary treatment combining a "cardio training" with muscle strengthening, supervised by qualified sports coaches, for a year, could reduce the impact of SA in the daily life of patients balanced by a biotherapy, compared to standard physiotherapy. This original care is part of the Adapted Physical Activity (APA), whose application decree came into force on March 1, 2017 and allows doctors to prescribe a physical therapy tailored to the needs of the patient. At present, the APA remains at the expense of the patients in ALD and in some cases, it can be supported, partially or totally, by the complementary health. APA could therefore be an alternative and / or complementary to physiotherapy as a physical therapy in the management of AS, in addition to pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 60 years old
* Present Axial Spondylitis meeting the criteria of ASAS 2009
* Be on treatment with biotherapy, stable dose for at least 6 months
* Complete the ALD criteria
* Have a BASFI score at inclusion ≤ 5
* Have signed the consent form
* Being able to be compliant to the study schedule (mobile and available)
* To be clinically stable for at least 6 months
* Affiliation to a social security scheme or beneficiary of such a scheme
* Does not present a contraindication to the practice of a physical activity

Exclusion Criteria:

* Regularly practice a sports activity (≥ 1hour / week)
* Have a severe handicap limiting the gestures of daily life (dressing, walking, etc ...)
* Have another significant osteo-articular pathology (Rheumatoid arthritis osteoarthritis, hip prosthesis ...)
* Have a bamboo column
* Being pregnant or planning to be pregnant in the coming year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-06-14 (Estimated)

PRIMARY OUTCOMES:
The mean variation of the BASFI score (Bath Ankylosing Spondylitis Functional Index) over a period of 18 months | 18 MONTHS
  The primary endpoint is the mean change in BASFI score (functional index of ankylosing spondylitis) between 12 months of management (or M12), and baseline (or M0), compared between the 2 groups. It will be noted BASFI (M12-M0). Patients follow-up will be done during 18 months.
  BASFI is a self-administered questionnaire that assesses the functional impact of the disease on the patient's life. This tool consists of 10 questions to answer a visual evaluation of 10 cm (0 for "easy" and 10 for "impossible").

SECONDARY OUTCOMES:
The mean variation of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 18 MONTHS
  This tool assesses disease activity based on the patient's response to 6 questions related to fatigue, joint and spinal joint pain, localized spot sensitivity, and morning stiffness (duration). and degree). Each answer can range from 0 (absent) to 10 cm (extreme) on a visual analogue scale or Likert scale. First, calculate the average for answers 5 and 6 and then calculate the average of the 5 values (the average value of answers 5 and 6 and the value of answers to the first 4 questions). It is a fast tool (with a filling time per patient from 30 seconds to 2 minutes), reliable and valid, also used for "routine" follow-up, at the request of the practitioner. This questionnaire is completed by the patient referring to his feelings during the last forty-eight hours.
The mean variation of C-reactive protein (CRP) and sedimentation rate (VS) over a period of 18 months | 18 MONTHS
  These 2 biomarkers of inflammation are regularly dosed as part of a "classical" follow-up by the rheumatologist, in addition to a more complete biological assessment. This assessment can be performed in the laboratory of biological analyzes of the choice of the patient. Patients follow-up will be done during 18 months.
  These values are retrieved at visits M0, M6, M12 and M18.
The mean variation of ASDAS (Ankylosing Spondylitis Disease Activity Score). | 18 MONTHS
  It is a new composite index to evaluate disease activity that combines 5 variables: 3 questions from BASDAI (2nd, 3rd and 6th), the value of CRP (or VS, if CRP not available ) and the EVA of the Global Assessment (EVA-AG) by the patient. This score has a good sensitivity and is calculated using the following formula:
  0.12 x Back Pain (0 to 10) + 0.06 x Duration of Morning Stiffness (from 0 to 10) + 0.11 x Patient Global (0 to 10) + 0.07 x Peripheral Bread / Swelling (0 to 10) + 0.58 x Ln (CRP (mg / l) +1)
The mean variation of the score of the Visual Analogue Scale of Global Appreciation (EVA-AG) over a period of 18 months. | 18 MONTHS
  The EVA-AG is a visual scale graduated from 0 (worst health condition imaginable) to 10 (best health imaginable) and the patient must indicate the appreciated value of his overall health condition on the scale and within a framework Reserve. Patients follow-up will be done during 18 months.
  The questionnaire is completed by the patient at each visit: M0, M6, M12 and M18.
The mean variation in NSAID consumption (Anti-Inflammatory Non Steroidal) over a period of 18 months. | 18 MONTHS
  The consumption of NSAIDs throughout the study is measured by completion by the physician of a questionnaire, based on the interview of the patient, which makes it possible to obtain the ASAS-NSAIDs (Assessment of SpondyloArthritis International Society - No Steroidal Anti-Inflammatory Drugs) score. It is calculated using a formula based on the daily dosage, the number of shots per week and the period of interest in days. Patients follow-up will be done during 18 months.
  This score is calculated at each visit over the 6 months preceding the visits: M0, M6, M12 and M18.
The mean variation in the consumption of analgesics. | 18 MONTHS
  The average consumption of analgesics, in the 6 months preceding the visit, is collected by the investigating doctor during the interrogation of the patient and transcribed in his medical file.
  Each treatment is informed as well as its daily dosage, the average number of days of weekly intake and the duration of it
The average variation in medical consumption over a period of 18 months | 18 MONTHS
  The medical consumption corresponds to the retranscription of all consultations, hospitalizations or other medical or paramedical care, in connection with his SA, carried out by the patient in the 6 months preceding the visit. Only non-research-related treatment consumptions are collected by the investigating physician and transcribed in his medical file. Physiotherapy sessions of the patient included in group 2, are not considered medical consumption, for example. Patients follow-up will be done during 18 months.
  This information is collected at each visit on the 6 months preceding the visits: M0, M6, M12 and M18.
Variation of items in the Patient Questionnaire. | 18 MONTHS
  The Patient Questionnaire is a questionnaire, to be completed by the patient, composed of 4 questions with 4 possible answers each time and a free commentary part.
  This questionnaire makes it possible to compare between the 2 groups, the adhesion and the satisfaction of the patients to their prescribed care and the frequency of realization of the recommended individual exercises, during the period of dedicated observation, as well as in follow-up.
The average change in scores on the Quality of Life Questionnaire (short form) SF-12. | 18 MONTHS
  The SF-12 is a self-questionnaire, non-pathology specific and can be administered to the general population, to assess the quality of life of the patient. This tool is an abbreviated version of the "Medical Outcomes Study Short-Form General Health Survey" (SF-36) with only 12 items out of 36, to assess the mental and physical health of the subject

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Joseph, Marseille, Bouches DU Rhone, France

IPD SHARING:
Plan to Share IPD: No